CLINICAL TRIAL: NCT04555772
Title: Evaluation of Factors That Cause Secondary Brain Damage on Mortality and Morbidity in Patients Undergoing Emergency Surgery Due to Head Trauma.
Status: Completed | Type: Observational
Sponsor: Turkish Society of Anesthesiology and Reanimation (Other)
Responsible Party: Sponsor
Other Study IDs: uludagunineuroanesthesia
Record Dates: First submitted 2020-07-29; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Brain Injuries
Keywords: secondary brain damage; electrolyte imbalance; head trauma
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Group: Patients who had been treated and recovered physically and gained cognitive functions completely.
  Interventions: Other: factors evaluation
- Sequel Group: Patients who could not gain their physical and cognitive functions.
  Interventions: Other: factors evaluation
- Exitus Group: Patients who did not respond to the treatments and lost their lives within 28 days of admission.
  Interventions: Other: factors evaluation

INTERVENTIONS:
Other: factors evaluation — They investigated mortality and morbidity in patients who underwent emergency operation within 24 hours after traumatic brain injury.

SUMMARY:
Traumatic brain injury is combination damage that occurs as a result of a chain reaction of various metabolic events that develop after primary damage caused by trauma. Pathological events such as lactic acidosis, electrolyte imbalance, increased inflammation that occur during traumatic brain injury leads to poor prognosis in patients.

The retrospective study was conducted to investigate the effect of factors that may cause secondary damage, especially electrolyte imbalance and blood glucose levels, on mortality and morbidity in patients undergoing emergency surgery due to head trauma.

ELIGIBILITY:
Inclusion Criteria:

* patients who admitted to Bursa Uludag University hospital between 2013 and 2018
* patients diagnosed with traumatic brain injury and operated within the first 24 hours after admission

Exclusion Criteria:

* pediatric patients
* patients that operated after 24 hour of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: they collect data of 108 patients who admitted to Bursa Uludag University hospital between 2013 and 2018 and were diagnosed with traumatic brain injury and operated within the first 24 hours after admission.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
mortality and morbidity in patients who underwent emergency operation within 24 hours after traumatic brain injury | 5 years
  It seems that secondary damage caused by metabolic events like eletrolyte imbalance in patients with head trauma should always keep in mind. If they encounter these situations, they should treat the patient and do replacements immediately.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa uludag university, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes